CLINICAL TRIAL: NCT06618196
Title: A Phase II, Randomized, Double-blind, Active-controlled, Parallel-group, Multicenter Study to Evaluate the Immunogenicity and Safety of DTaP-HepB-IPV-Hib Hexavalent Vaccine LR20062 Versus Hexaxim Administered Intramuscularly in Healthy Infants As Primary Series At 2, 4, 6 Months of Age
Brief Title: Study to Evaluate the Immunogenicity of LR20062 Compared to Control When Administered Intramuscularly in Healthy Infants At 2, 4, 6 Months of Age
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LG-VGCL002
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis; Haemophilus Influenzae Type B Infection
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Haemophilus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Any persons accompanying the subject for the site visits, including parents, other family members, and/or legally acceptable representatives, will be shielded from view by physical barriers while the study vaccine is administered. The unblinded site personnel for the preparation/administration of study vaccines will keep the unblinded information separate from those persons for any study related procedures/assessments after administration of study vaccines, which includes all safety follow-up procedures. Blinded site personnel will be responsible for all safety and immunogenicity follow-up procedures after study vaccine administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Test group 1 (Experimental): Low dose of candidate hexavalent vaccine (DTaP-HepB-IPV-Hib)
  Interventions: Biological: LR20062
- Test group 2 (Experimental): Middle dose of candidate hexavalent vaccine (DTaP-HepB-IPV-Hib)
  Interventions: Biological: LR20062
- Test group 3 (Experimental): High dose of candidate hexavalent vaccine (DTaP-HepB-IPV-Hib)
  Interventions: Biological: LR20062
- Test group 4 (Active Comparator): Control hexavalent vaccine (DTaP-HepB-IPV-Hib)
  Interventions: Biological: DTaP-HepB-IPV-Hib vaccine

INTERVENTIONS:
Biological: LR20062 — DTaP-HepB-IPV-Hib vaccine
  Arms: Test group 1; Test group 2; Test group 3
Biological: DTaP-HepB-IPV-Hib vaccine — Control hexavalent vaccine
  Arms: Test group 4

SUMMARY:
This is a phase II, randomized, double-blind, active-controlled, parallel-group, multicenter study to evaluate the immunogenicity and safety of DTaP-HepB-IPV-Hib hexavalent vaccine LR20062 in healthy infants as primary series at 2, 4, 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female aged two months (50 to 70 days inclusive) on the day of the first dose of study vaccine.
2. Is born at full term of pregnancy (≥37 weeks of gestation) with a birth weight of ≥2.5 kg.

Exclusion Criteria:

Medical conditions:

1. Has a history of diphtheria, tetanus, pertussis, poliovirus, Hep B, or Hib infection.
2. Has a known SARS-CoV-2 infection at Screening.
3. Was born to a mother with a known history of Hep B infection based on HBsAg seropositivity.
4. Was born to a mother with a known history of HIV infection based on HIV antibody seropositivity.
5. Had a recent febrile illness, defined as axillary temperature ≥38.0℃ [≥100.4℉] occurring at or within 72 hours prior to receipt of study vaccine.

   Prior/concomitant therapy:
6. Has previously received vaccination against diphtheria, tetanus, pertussis, poliovirus, and/or Hib infections since birth.
7. Has received or is expected to receive immunosuppressive agents or other immune-modifying drugs during the conduct of the study.
8. Meets one or more of the following systemic corticosteroid exclusion criteria:

   1. Has received systemic corticosteroids (equivalent of ≥0.5 mg/kg total daily dose of prednisone) for ≥14 consecutive days and has not completed treatment at least 30 days prior to Screening.
   2. Is expected to require any systemic corticosteroids during conduct of the study.

   Note: Topical, ophthalmic, and inhaled steroids are permitted at the discretion of the Investigator.
9. Has received any non-study vaccine within 30 days before the first dose of study vaccine or is scheduled to receive any other vaccine within one month after the third dose of study vaccine.

Exception: Vaccines against BCG and Hep B at birth, rotavirus, MMR, and PCV if received according to the routine immunization schedule, and inactivated influenza vaccine, are allowed.

Ages: 50 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 336 (Estimated)
Dates: Start 2024-10-02 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Seroprotection/vaccine-response rate | 1 month after the third dose primary series
  * Proportion of subjects achieving seroprotection to each antigenic components
  * Proportion of subjects with vaccine response for pertussis antigens

SECONDARY OUTCOMES:
Geometric mean concentration (GMC) or Geometric mean titer (GMT) | 1 month after the third dose primary series
  GMC or GMT and their ratio of all types of antibodies
Seroconversion rate | 1 month after the third dose primary series
  Proportion of subjects achieving seroconversion to pertussis and poliovirus
Long-term seroprotection rate | 1 month after the third dose primary series
  Proportion of subjects with seroconversion for diphtheria, tetanus, and Hib antigens
Solicited adverse event | 7 days after each vaccination
  Expected local or systemic side effects after vaccination
Unsolicited adverse event | 1 month after each vaccinations
  Any AEs other than solicited AEs
Immediate reactions after vaccination | 30 minutes after each vaccination
  Any AEs that occur within 30 minutes after the study vaccine administration